CLINICAL TRIAL: NCT07186062
Title: Clinical Outcomes of Levosimendan Versus Dobutamine Versus Milrinone in Cases With Acute Decompensated Heart Failure With Impaired Renal Function
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Khaled Abdou, assistant professor, Ain Shams University
Other Study IDs: FMASU MD 185a/2022/2023
Record Dates: First submitted 2025-09-10; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Acute Decompensated Heart Failure (ADHF); Cardiorenal Syndrome (CRS)
Keywords: Levosimendan; dobutamine; Milrinone; Acute Decompensated Heart Failure (ADHF); Cardiorenal Syndrome (CRS)
MeSH Terms: conditions — Cardio-Renal Syndrome | interventions — Simendan; Dobutamine; Milrinone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Levosimendan group
  Interventions: Drug: Levosimendan
- Dobutamine group
  Interventions: Drug: Dobutamine
- Milrinone group
  Interventions: Drug: Milrinone

INTERVENTIONS:
Drug: Levosimendan — Inotropic agents titrated to response to keep mean arterial blood pressure above 55 mmHg :
  •Levosimendan: loading dose 6-12 microgram/ kg then continuous infusion of 0.05-0.2 µg/kg/min.
  Groups: Levosimendan group
Drug: Dobutamine — Inotropic agents titrated to response to keep mean arterial blood pressure above 55 mmHg :
  • Dobutamine: continuous infusion starting at 2.5 µg/kg/min, titrated up to 20 µg/kg/min as needed.
  Groups: Dobutamine group
Drug: Milrinone — Inotropic agents titrated to response to keep mean arterial blood pressure above 55 mmHg :
  • Milrinone: 50 mcg/kg loading dose, then 0.375-0.75 mcg/kg/min IV according to patient response.
  Groups: Milrinone group

SUMMARY:
This study aimed to assess and compare the cardiac, renal, and clinical efficacy of Levosimendan (LEV), Dobutamine (DOB), and milrinone (MIL) in cases with acute decompensated heart failure (ADHF) complicated by renal impairment, with a focus on their role in the management of cardiorenal syndrome (CRS).

DETAILED DESCRIPTION:
Methods Upon ICU admission and once the clinical decision to initiate inotropic therapy was made, all enrolled patients underwent a standardized evaluation protocol that included: Comprehensive medical history and clinical examination. Laboratory assessments, including Complete blood count (CBC), Arterial blood gases (ABG), Liver and kidney function tests, Serum electrolytes, Random blood glucose, Estimated glomerular filtration rate (eGFR). Cardiac parameters were recorded by EV1000 clinical platform device to assess the cardiac index (CI), stroke volume variations (SVV), and systemic vascular resistance index (SVRI). at baseline, 24 hours after inotropic therapy initiation, and again on day 7 or prior to ICU discharge whichever occurred first. Renal function indicators _including serum creatinine, blood urea nitrogen (BUN), eGFR, and urinary output_ were measured before the start of infusion and monitored daily until ICU discharge or death.

Medications were routinely administered as part of standard institutional practice. Where trial-specific medications were used, we have provided a clear distinction between these and routine medications. omission of medications not routinely used in our protocol did not cause harm to patients, and all treatments provided were in accordance with current safety standards and ethical guidelines.

Inotropic agents titrated to response to keep mean arterial blood pressure above 55 mmHg :

* Levosimendan: loading dose 6-12 microgram/ kg then continuous infusion of 0.05-0.2 µg/kg/min.
* Dobutamine: continuous infusion starting at 2.5 µg/kg/min, titrated up to 20 µg/kg/min as needed.
* Milrinone: 50 mcg/kg loading dose, then 0.375-0.75 mcg/kg/min IV according to patient response.

Primary outcomes included changes in cardiac and renal function parameters. Pre- and post-infusion values were compared to assess treatment response.

Secondary outcomes encompassed length of ICU stay, total hospital stay, ICU readmission, and all-cause in-hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years old) patients with ADHF (LVEF ≤ 40% documented prior to enrollment) admitted to the ICU with renal impairment (estimated GFR between 30 and 60 mL/min/1.73 m², calculated using the Modification of Diet in Renal Disease Study equation (MDRD equation)) and require inotropic support.

Exclusion Criteria:

Cases were excluded from the study if they met any of the following criteria:

* Age younger than 18 years
* Untreated acute HF
* Resting heart rate exceeding 120 beats per minute
* Recent MI or acute coronary syndrome within the previous two months
* Diagnosed pulmonary embolism
* Structural cardiac conditions
* Known history of kidney disease diagnosed prior to HF
* Administration of contrast agents or nephrotoxic drugs within the previous seven days
* Severe liver dysfunction (Child C)
* Active acute inflammatory or infectious diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (>18 years old) patients with ADHF (LVEF ≤ 40% documented prior to enrollment) admitted to the ICU with renal impairment (estimated GFR between 30 and 60 mL/min/1.73 m², calculated using the Modification of Diet in Renal Disease Study equation (MDRD equation) [10] and require inotropic support.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
renal function parameters. | 7 days
  Changes in serum creatinine (mg/dl). Pre- and post-infusion values were compared to assess treatment response.
renal function | 7 days
  Changes in serum BUN (mg/dl). Pre- and post-infusion values were compared to assess treatment response.
renal function | 7 days
  Changes in eGFR (mL/min/1.73 m²). Pre- and post-infusion values were compared to assess treatment response.
renal function | 7 days
  Changes in urine output (mL/day). Pre- and post-infusion values were compared to assess treatment response.
cardiac function | 7 days
  changes in ejection fraction % by transthoracic echocardiography. Pre- and post-infusion values were compared to assess treatment response.
cardiac function | 7 days
  Changes in cardiac index (L/min/m²) measured by EV1000 clinical platform device. Pre- and post-infusion values were compared to assess treatment response.
cardiac function | 7 days
  changes in stroke volume variations (SVV) measured by EV1000 clinical platform. Pre- and post-infusion values were compared to assess treatment response.
cardiac function | 7 days
  changes in systemic vascular resistance index (SVRI) using EV1000 clinical platform device. Pre- and post-infusion values were compared to assess treatment response.

SECONDARY OUTCOMES:
morbidity | 28 day
  length of ICU stay (days).
morbidity | 28 day
  Total hospital stay (days)
morbidity | 28 day
  ICU readmission
mortality | 28 day
  In-hospital mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine Ain shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided